CLINICAL TRIAL: NCT06737900
Title: Effects Of Jandas Approach Versus Proprioceptive Neuromuscular Facilitation Technique On Pain, Range of Motion, Disability, Endurance And Quality Of Life In Patients With Lower Cross Syndrome
Brief Title: Effects Of Jandas Approach Vs PNF Technique On Pain, ROM, Disability, Endurance And QOL In Patients With LCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0107
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Lower Cross Syndrome
Keywords: Disability, Muscle strength, Pain, Quality of life, range of motion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: there were total of 52 participants and were randomly assigned to two different groups. Group A received proprioceptive neuromuscular facilitation technique and Group B received jandas approach of stretching and strengthening.
  The aim of this study was to study the Effects of Jandas approach versus Proprioceptive Neuromuscular Facilitation technique on pain, disability, range of motion, endurance and quality of life in patients with lower crossed syndrome
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional physical therapy (Active Comparator): Heating pad for 10 minutes and Core stability exercises for 20 minutes with 10 seconds of rest intervals.
  Interventions: Other: jandas approach
- Proprioceptive Neuromuscular Facilitation technique (Experimental): Heating pad for 10 minutes and core stability exercises for 20 minutes along with Proprioceptive Neuromuscular Facilitation technique was used for stretching and rhythmic stabilization technique for strengthening. Stretching was performed using contract-relax technique.
  Interventions: Other: traditional physical therapy

INTERVENTIONS:
Other: traditional physical therapy — * Heating pad for 10 minutes
  * Core stability exercises for 20 minutes with 10 seconds of rest intervals
  * Patients were advised to stretch for 5 minutes then perform lumber stability exercises.
  * These stability exercises included side bridges, supine extension bridge, straight leg raise in prone lying, alternate arm and leg raise from quadruped position and prone bridges.
  Both groups took sessions thrice a week for a total of 4 weeks.
  Arms: Proprioceptive Neuromuscular Facilitation technique
Other: jandas approach — * Stretching exercise for erector spinae and back extensors muscles
  * Stretching exercises for iliopsoas muscle and rectus femoris muscle
  * Strengthening exercise for abdominal muscle and gluteal maximus muscle Stretching exercise was performed actively for 3 repetitions x 1 set and 4 days a week Strengthening exercise was performed for 10 second hold and 10 repetitions. All Exercises was performed 3 times per week for total of 4 weeks
  Arms: traditional physical therapy

SUMMARY:
The goal of this randomized clinical trial is to learn if the given interventions that is jandas approach versus Proprioceptive Neuromuscular Facilitation technique can treat pain, disability, range of motion, endurance and quality of life in patients with Lower cross syndrome on both genders and age group of 25-40 years. The main questions it aims to answer are:

Does jandas approach versus Proprioceptive neuromuscular facilitation technique improves pain, disability, range of motion, endurance and quality of life in patients with lower cross syndrome?

There is a comparison between two groups: Researchers will compare the jandas approach and proprioceptive neuromuscular facilitation technique to see if there is effects on pain, disability, range of motion, endurance and quality of life in patients with lower cross syndrome.

Participants in group A will be given

* Heating pad for 10 minutes
* Core stability exercises for 20 minutes with 10 seconds of rest intervals
* Proprioceptive Neuromuscular Facilitation technique was used for stretching of erector spinae, quadratus lumborum, rectus femoris and iliopsoas and rhythmic stabilization technique for strengthening. Stretching was performed using contract-relax technique in supine, prone and side lying positions. The Contract-Relax method included the target muscle to be lengthened and held in lengthened position while the patient contracted the Target-Muscle to its maximum position isometrically 3 to 6 seconds.
* Rhythmic stabilization technique was used to strengthen and stabilize the postural trunk muscles of hip: Abdominals and gluteal muscles strengthening and Participants in group B will be given
* Heating pad for 10 minutes
* Core stability exercises for another 20 minutes.
* After which it was treated with the Janda's approach of musculoskeletal pain that includes strengthening of the weakened muscles and stretching of the tightened muscles including Stretching exercise for erector spinae and back extensors muscles Stretching exercises for iliopsoas muscle and rectus femoris muscle Strengthening exercise for abdominal muscle and gluteal maximus muscle

DETAILED DESCRIPTION:
A Randomized Clinical Trial was conducted at Riphah Clinic Lahore. A total of 52 patients (N=52) were assessed for eligibility criteria through non-probability consecutive sampling technique. 6 participants were excluded from the research. These 6 patients rejected to be the part of the study and declined any treatment. Hence 46 participants were included in the study that were first assessed and diagnosed with lower cross syndrome and met the inclusion criteria. As a result, total of 46 patients including (females: 39, males: 7) were considered eligible for the study. They were randomized through computer generated software. The list was concealed by a sealed envelope. The group A was labeled as 1 and group B was labeled as 2. Patients enrolled in this study have age between 25-40 years. Consent form was filled before the start of the treatment. The participants were randomly enrolled into two groups named as group A and group B. Baseline assessment of pain, disability, quality of life, lumbar range of motion, hip range of motion and endurance was taken using NPRS, ODI, SF-36, inclinometer, goniometer and McGill test of endurance respectively, before the start of the treatment by an assessor. Both groups: A and B received baseline treatment that consisted of a heating pad for 10 minutes followed by core stability exercises for 20 minutes with 10 seconds of rest intervals. Patients were advised to stretch for 5 minutes then perform lumber stability exercises.

Group A The group A first received the baseline treatment mentioned above then Proprioceptive Neuromuscular Facilitation technique for stretching and rhythmic stabilization technique for strengthening. PNF stretching was performed using contract-relax technique in supine, prone and side lying positions. The Contract-Relax method includes the target muscle to be lengthened and held in lengthened position while the patient will contract the Target-Muscle to its maximum position isometrically for an allotted amount of time that varies from 3 to 6 seconds. The muscle which is contracting is the agonist and the muscle which is relaxing is called the antagonist.

• Erector spinae stretching: Ask the patient to lie down and bring both the legs up to their chest by grabbing around their knees to stretch erector spinae muscle. Ask the patient to tuck in their chin and hold the stretch for 6 seconds of contraction with 80% force of the maximal isometric contraction on the erector spinae followed by a 15-second passive static stretching in the opposite direction of the muscle.

Quadratus lumborum stretching: the patient will perform active lateral flexion of the spine. To stretch the right QL the patient will laterally flex the spine to the left and vice versa. Ask the patient to hold the lateral flexion for 6 seconds of contraction with 80% force on the of the maximal isometric contraction on the muscle followed by a 15-second passive static stretching in the opposite direction of the muscle.

Rectus femoris stretching: the patient will lie in a side lying position on the treatment couch. The patient will flex the uppermost testing knee backwards and the therapist will hold onto above the foot of the patient, bend the knee to 90 degree and will pull the hip into extension and will ask the patient to hold a 6 second contraction with 80% force of the maximal isometric contraction of muscle followed by a 15-second passive static stretching in the opposite direction of the muscle.

Iliopsoas stretching: by using the modified Thomas test position, the patient will lie supine on the treatment table. Ask the patient to hold the unaffected leg towards their chest, the therapist will then hold the leg to be stretched above the knee and will provide a constant force to stretch and extend the leg. The contractions will be held for 6 seconds with 80% force of the maximal isometric contraction of muscle followed by a 15-second passive static stretching in the opposite direction of the muscle Rhythmic stabilization technique; is also a PNF technique that is shown to strengthen and stabilize the postural trunk muscles of hip and shoulder girdle. Therefore it will be used for the strengthening of the abdominal muscles and the gluteal muscles.

• Abdominals and gluteal muscles strengthening: Ask the patient to lie on the mat with both the knees flexed. The patient will raise their hips and perform a glute hold for 2 to 5 seconds against the resistance applied by the therapist. Hip rolls can also be performed by the patient in each direction against the resistance applied by the therapist.

Group B: The group B received heating pad for 10 minutes and core stability exercises for another 20 minutes after which it was treated with the Janda's approach of musculoskeletal pain that includes strengthening of the weakened muscles and stretching of the tightened muscles. This approach included:

* Stretching exercise for erector spinae and back extensors muscles
* Stretching exercises for iliopsoas muscle and rectus femoris muscle
* Strengthening exercise for abdominal muscle and gluteal maximus muscle. Stretching exercise will be performed actively for 30 second hold and 3 repetitions.

Strengthening exercise will be performed for 10 second hold and 10 repetitions. All Exercise will be performed 3 times per week for total of 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age group of 25-40 years.
* Both genders male and female.
* NPRS score range from 4-7.
* Modified Thomas test positive , Back extensor test positive, prone hip extension strength test positive , Trunk flexion strength test positive.

Exclusion Criteria:

* Vertebral Fractures
* Tumors
* Pregnancy
* Diagnosed psychological disorders

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
numerical pain rating scale | 4th day
  changes from baseline numerical pain rating scale is a scale that was used to measure pain of the patient and ranges from 0 to 10. 0 gives an indication of no pain and 10 gives an indication of worst pain.
owestry disability index | 4th day
  changes from baseline in functional impairment and disability, Owestry Disability Index was used. ODI consist of 10 items that are related to daily living activities limitation with 6 levels being set in each dimension. The score of 0 indicates the disability of lowest level, while 5 is an indication of disability of highest level. The overall score is then converted in percentage out of 100%

SECONDARY OUTCOMES:
SF-36 | 4th day
  Changes from baseline sf-36 was used to assess the quality of life. it consists of 8 domains covering physical and mental health. norm based scoring system is used with a mean of 50 ad standard deviation of 10. scores above 50 indicated a better health related quality and below 50 suggest below average health.
ROM lumber spine (flexion) | 4th day
  changes from baseline lumber flexion range of motion was assessed by inclinometer
ROM lumber spine (extension) | 4th day
  changes from baseline in lumber spine extension range of motion was assessed through inclinometer
ROM lumber spine (lumber right lateral flexion) | 4th day
  changes from baseline in lumber right lateral flexion range of motion was assessed through inclinometer
ROM lumber spine (lumber left lateral flexion) | 4th day
  changes from baseline in lumber left lateral flexion range of motion was assessed through inclinometer
ROM hip (flexion) | 4th day
  changes from baseline in hip flexion range of motion was assessed through a goniometer
ROM hip (extension) | 4th day
  changes from baseline in hip extension range of motion was assessed through a goniometer
McGill trunk flexion endurance | 4th day
  changes from baseline in trunk flexion endurance was assessed by The McGill Torso Endurance Test. these are a useful battery of tests that assess all sides of the trunk allowing us to assess the endurance capacity of the torso muscles or if there is an imbalance between the muscle groups which can contribute to low-back dysfunction and core instability
McGill trunk extension endurance | 4th day
  changes from baseline in trunk extension endurance was assessed by The McGill Torso Endurance Test. these are a useful battery of tests that assess all sides of the trunk allowing us to assess the endurance capacity of the torso muscles or if there is an imbalance between the muscle groups which can contribute to low-back dysfunction and core instability
McGill trunk right lateral endurance | 4th day
  changes from baseline in trunk right lateral endurance was assessed by The McGill Torso Endurance Test. these are a useful battery of tests that assess all sides of the trunk allowing us to assess the endurance capacity of the torso muscles or if there is an imbalance between the muscle groups which can contribute to low-back dysfunction and core instability
McGill trunk left lateral endurance | 4th day
  changes from baseline in trunk left lateral endurance was assessed by The McGill Torso Endurance Test. these are a useful battery of tests that assess all sides of the trunk allowing us to assess the endurance capacity of the torso muscles or if there is an imbalance between the muscle groups which can contribute to low-back dysfunction and core instability

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehab Training and Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1) authors: rajalaxmi v, nandhini g etc, article name: efficacy of jandas approach versus brueggers exercise in pelvic cross syndrome and its impact on quality of life, journal name: JK welfare and pharmascope foundation, publication date: 8 feb 2020, volume and pages were not mentioned